CLINICAL TRIAL: NCT01345396
Title: Assessment of an Educational Programme for Pregnant Asthmatic Women on the Level of Asthma Control and Unscheduled Doctor Visits During the Pregnancy
Brief Title: Influence of an Asthma Education Programme on Asthma Control During Pregnancy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Vincent Ninane, Prof. Dr. V. Ninane, Centre Hospitalier Universitaire Saint Pierre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B07620096465
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Asthma
Keywords: Asthma; Health education; Pregnancy
MeSH Terms: conditions — Asthma; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education (Experimental)
  Interventions: Behavioral: Health education about asthma
- No education (No Intervention)

INTERVENTIONS:
Behavioral: Health education about asthma — Three face-to-face appointments (<20, 36 weeks of gestation and 12 weeks after the baby birth). Topics: What is asthma? What influence the course of asthma? How to monitor it? How to manage it?
  Arms: Education

SUMMARY:
Asthma is the most frequent respiratory disease during pregnancy. In a third of cases, the level of asthma control can decrease during the pregnancy, especially between the 29th and the 36th week. The occurrence of such complications are linked with a high asthma severity level just before the conception and an history of respiratory complications in a previous pregnancy. Many reviews and recommendations claim that pregnant women with asthma should be included in an educational progamme. However, this is poorly studied. The purpose of this study is to observe if an educational programme given before the 20th weeks of gestation has an effect on asthma control until the end of gestation.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman (less than 20 weeks of gestation at the inclusion time)
* Diagnosis of asthma before the pregnancy (clinical history and specific medications used)
* Agreement to enter into the study

Exclusion Criteria:

* Pregnant woman (more than 20 weeks of gestation at the inclusion time)
* History of major respiratory problems during previous pregnancy(ies)
* Refusal to enter into the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-02 (Actual); Study Completion 2015-12

PRIMARY OUTCOMES:
The level of asthma control | Inclusion (baseline), 36 weeks of gestation, 12 weeks post partum
  Assessment by the Asthma Control Questionnaire

SECONDARY OUTCOMES:
Number of unscheduled visits to the doctor for asthma | Inclusion (baseline), 36 weeks of gestation, 12 weeks post partum
Quality of life | Inclusion (baseline), 36 weeks of gestation, 12 weeks post partum
  Asthma Quality of life questionnaire
Knowledge about asthma | Inclusion (baseline), 36 weeks of gestation, 12 weeks post partum
  Survey of asthma knowledge of French language Questionnaire de connaissance de l'asthme de langue française

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ninane, MD PhD, Principal Investigator — CHU St Pierre Brussels
Locations (1):
- CHU St Pierre; pulmonology department, Brussels, Belgium